CLINICAL TRIAL: NCT03593148
Title: The Effect of Lifestyle Treatment on Physical Capacity, Maximal Strength, Eating Behavior and Quality of Life in Patients With Morbid Obesity
Brief Title: The Effect of Lifestyle Treatment in Patients With Morbid Obesity
Acronym: LIFETIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: University college of south-east Norway (Unknown)
Responsible Party: Principal Investigator, Jarle Berge, Principal investigator, Sykehuset i Vestfold HF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIFETIME
Record Dates: First submitted 2018-04-30; First posted 2018-07-19 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Physical Capacity; Leg Strength; Eating Behavior; Life of Quality
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle treatment (Other): Patients will be included in the Lifestyle treatment that is a existing treatment program at Vestfold Hospital Trust.
  Interventions: Other: Lifestyle

INTERVENTIONS:
Other: Lifestyle — Lifestyle treatment

SUMMARY:
The effect of lifestyle treatment on physical capacity, maximal strength, eating behavior and quality of life in patients with morbid obesity (LIFETIME)

DETAILED DESCRIPTION:
In this study, the investigators will investigate whether more intensive day-based lifestyle treatment process have a better effect on weight loss and health-related quality of life than a previous treatment. Investigators also want to investigate whether patients with good physical capacity (maximal oxygen uptake) and bone strength (maximum bone strength) before initiating treatment and / or after 3 and 6 months intensive training may have greater weight loss 1 and 2 years after treatment than patients with lower physical capacity and bone strength.

ELIGIBILITY:
Inclusion Criteria:

* Treatment seeking morbidly obese patients (BMI ≥ 40 kg/m2 or BMI 35 to 39.9 kg/m2 with ≥ 1 co morbidity) attending the Vestfold Hospital Trust.

Exclusion Criteria:

* Uncompensated heart failure
* Recent myocardial infarction or stroke (<½ years)
* Severe arrhythmia or heart failure
* Unstable angina pectoris
* Renal failure
* Pregnancy
* Severe eating disorders
* Active substance abuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Weight change at 2-year follow up | Changes from baseline body weight at 2-year follow up.
  Effect of intensive treatment on weight loss changes at 2- year follow up.
  Body weight was measured with patients wearing light clothing and no shoes on Scanvaegt DS-530 (Århus, Denmark) at baseline and at 2-year follow up.

SECONDARY OUTCOMES:
Maximal leg strength change at 2-year follow up | Changes from baseline maximal leg strenght at 2-year follow up.
  Maximum leg strength will be measure with a bone press device (OPS161 Interchangeable Leg Press) at baseline, after 3-6 month and 1-2 years. The test will be conduct as an individual adapted protocol with gradual loading until voluntary maximum bone strength is achieve.
Physical capacity change at 2-year follow up | Changes from baseline physical capacity at 2-year follow up.
  Physical capacity will be measure as maximum oxygen uptake (VO2max) by indirect calorimetry (Jaeger Oxycone Pro) at baseline, after 3-6 month and 1-2 years. Indirect calorimetry is to be regard as a gold standard for measurement of maximum oxygen uptake.
Health-related quality of life (HRQoL) - Short Form Health Survey (RAND-36), change at 2-year follow up | Changes from baseline RAND-36 at 2-year follow up.
  The patient reported outcome measurements (PROMS) comprise three elements; generic and obesity specific health related quality of life (HRQoL) and obesity specific symptoms measured at baseline, 3 months, 6 months, 1 year and 2 years.
  The RAND-36 is a 36-item measure of generic HRQOL consisting of eight additive subscales (Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health) and two summary scores each based on four subscales (Physical Component Summary and Mental Component Summary). Scores on all subscales range from 0 to 100. Summary-scores will be norm-based, with mean (SD) 50 (10). Higher scores on all scales represent better HRQOL.
Health-related quality of life (HRQoL) - Impact on Weight Questionnaire (IWQOL-Lite), change at 2-year follow up | Changes from baseline IWQOL-Lite at 2-year follow up.
  The patient reported outcome measurements (PROMS) comprise three elements; generic and obesity specific health related quality of life (HRQoL) and obesity specific symptoms measured at baseline, 3 months, 6 months, 1 year and 2 years.
  The IWQOL-Lite is a 31-item measure of weight-related quality of life. There are five domain scores (Physical Function, Self-Esteem, Sexual Life, Public Distress and Work) and a total score. Scores for all domains and total score range from 0-100, with lower scores indicating greater impairment.
Health-related quality of life (HRQoL) - Weight-Related Symptom Measure (WRSM), change at 2-year follow up | Changes from baseline WRSM at 2-year follow up.
  The patient reported outcome measurements (PROMS) comprise three elements; generic and obesity specific health related quality of life (HRQoL) and obesity specific symptoms measured at baseline, 3 months, 6 months, 1 year and 2 years.
  The WRSM is a 20-item measure for the presence and distress of 20 weight-related symptoms. The distress scores of the symptoms are reported on a six-point likert scale. Two summary scores are calculated; an additive score of presence of symptoms ranging from 1 to 20 and a symptom distress score for all symptoms. Symptom distress scores range from 0 to 100, with higher scores indicating a higher or worse total symptom distress.
Binge Eating Scale (BES), change at 2-year follow up | Changes from baseline BES at 2-year follow up.
  The patient reported outcome measurements (PROMS) eating behavior at baseline, 3 months, 6 months, 1 year and 2 years.
  The Binge Eating Scale comprise 16 items assessing binge eating problems. Additive scores range between 0-46, with higher scores indicating greater problems. Cut-off scores have been established to determine binge severity, with "severe" represented by scores > 27, "moderate" by scores 18-26, and "mild-none" by scores < 17.
The Power of Food scale (PFS) change at 2-year follow up | Changes from baseline PES at 2-year follow up.
  The patient reported outcome measurements (PROMS) eating behavior at baseline, 3 months, 6 months, 1 year and 2 years.
  The Power of Food scale assess both the psychological impact and respondent's responsiveness to a food-abundant environment. This is a 15-item scale whose items pertain to three situations: food being readily available in the environment but not physically present, food is physically present, but not tasted, and food is first tasted but not already consumed. The three subscales is scored 0-100 with higher scores indicating greater eating problems.
Weight change at 1-year follow up | Changes from baseline body weight at 1-year follow up.
  Effect of intensive treatment on weight loss changes after 1- year follow up
  Body weight was measured with patients wearing light clothing and no shoes on Scanvaegt DS-530 (Århus, Denmark) at baseline and at 1-year follow up.
Three Factor Eating Questionnaire (TFEQ - R21) | Changes from baseline TFEQ-R21 at 2-year follow up.
  The patient reported outcome measurements (PROMS) eating behavior at baseline, 3 months, 6 months, 1 year and 2 years.
  TFEQ-R21 consists of 21 questions that measure cognitive and emotional conditions related to food intake, as well as degree of control over food intake. Each item scores either 0 or 1 point.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hertel, PhD, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Jarle Berge, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03593148/Prot_SAP_000.pdf